CLINICAL TRIAL: NCT03468881
Title: Development and Feasibility of a Communication Training Package for Therapeutic Radiographers to Manage Emotional Talk With Breast Cancer Patients in Treatment
Brief Title: A Communication Skills Package to Prevent Fear of Cancer Recurrence
Acronym: FORECAST2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of St Andrews (Other)
Collaborators: NHS Lothian (Other Government); Breast Cancer Now (Other)
Responsible Party: Principal Investigator, Prof G Humphris, Chair of Health Psychology, University of St Andrews
Other Study IDs: 2017MayPR898
Record Dates: First submitted 2018-02-20; First posted 2018-03-19 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer radiation therapy: Observation over a period of all treatment sessions for radiotherapy.
  Interventions: Other: Communication Skills Training Package (KEW)

INTERVENTIONS:
Other: Communication Skills Training Package (KEW) — A training package (called KEW: Know, Encourage and Warm-up) for therapeutic radiographers to manage emotional talk with breast cancer patients in treatment.

SUMMARY:
This study (FORECAST 2) builds upon the work of the successful pilot study (FORECAST) that found some evidence that breast cancer patients' fears of cancer recurrence (FCR) were sensitive to the communication exchange with therapeutic radiographers during weekly review appointments. The aim of FORECAST 2 is to co-design and pilot a communication training package for therapeutic radiographers to help them manage emotional talk with breast cancer patients who are undergoing treatment, with the intention to minimise patients' development of FCR during this trajectory.

DETAILED DESCRIPTION:
The first aim of this study is to develop a training package (called KEW: Know, Encourage and Warm-up) to enhance communication skills of therapeutic radiographers in responding to emotions and concerns that are expressed by breast cancer patients at weekly review appointments. The first two phases of the project address this aim. Phase 1 will use a co-design methodology in which patients and therapeutic radiographers come together to develop a storyboard for the video and manual that will comprise the training package. Both local and national patient representatives and radiographers will be asked to comment and provide feedback on the output of the co-design process, leading to the production of the training video and manual (phase 2). Data collection will include verbatim transcripts from the co-design process, which will be content analysed to identify recommended techniques to be used within the review radiotherapy setting.

Phase 3 of the project addresses the second study aim, which is to pilot the package in a single service to test the acceptability into routine practice, to collect details for the preparation of a RCT study that includes more service units, to produce an electronic diary assessment of recurrence fears and to observe practice benefits within service. A pilot workshop will be conducted, after which 74 (female) breast cancer patients will be recruited to participate. All measures required for the RCT will be included.

Patients will complete questions including: 1) demographic information, 2) a 7-item FCR scale (FCR7) and 3) a 20-item Affect Schedule (PANAS) before first radiation treatment (T1). Throughout the period of treatment, patients will be asked to fill in a daily 3-item FCR questionnaire (FCR3) either in the form of a paper dairy or through a mobile phone application to monitor their FCR level. Then, at the end of the radiotherapy treatment (T2), PANAS and FCR7 will be measured again. Patients will also be asked to complete an adaptation of the Medical Interview Satisfaction Sale (MISS) and the Consultation and Relational Empathy measure (CARE). Finally, six-eight weeks after the end of the treatment (T3), all participants will be asked to complete the FCR7 once again as well as a 5-item EuroQoL EQ-5D-3L scale by telephone.

The same system of latent variable growth curve analysis as in the pilot FORECAST study will be used to calculate patients' FCR trajectory and link these to FCR7 outcomes. With a sample size of 74 patients, a medium to low-sized effect of 0.375 at 80% power and alpha (2-sided) set to 0.05 can be detected to demonstrate if the KEW intervention can decrease levels of FCR compared to the FCR levels obtained in the FORECAST pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who are diagnosed with breast cancer, age 18+

Exclusion Criteria:

* Under 18 years old
* Male
* Known psychiatric illness
* Receiving palliative radiotherapy (non-curative)
* Unable to communicate in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To evaluate the co-designed communication training package, 74 breast cancer patients receiving radiotherapy at the Edinburgh Cancer Centre will be recruited.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Fear of Recurrence level - FCR7 | 6-8 weeks after treatment
  The Fear of Recurrence level scale (FCR7) is a 7-item self-report measure of patients' fear of cancer recurrence. It has been used previously in a national study and the FORECAST pilot. It shows high internal consistency (Cronbach's α of 0.92) and its construct validity has been demonstrated through association with the Hospital Anxiety and Depression Scale (HADS) (Humphris et al., 2018).

SECONDARY OUTCOMES:
Fear of Recurrence level - FCR3 | up to 4 weeks from baseline visit
  The Fear of Recurrence level scale (FCR3) is a 3-item self-report measure of patients' fear of cancer recurrence. It has been used previously in the FORECAST pilot study and is based on the 4-item scale FCR4, which psychometric qualities are supportive of its internal consistency (Cronbach's α of 0.92) and validity (association with the Hospital Anxiety and Depression Scale (HADS)) (Humphris et al., 2018).
Positive And Negative Affect Schedule (PANAS) | 4 weeks following baseline visit
  The Positive and Negative Affect Schedule (PANAS) is a 20-item self-report measure of positive and negative affect. The PANAS has been shown to possess adequate psychometric properties in a large sample drawn from the general adult population, and the construct validity of the PANAS scales and the reliabilities of both scales were adequate, Cronbach's α were 0.89 for Positive Affectivity and 0.85 for Negative Affectivity (Crawford & Henry, 2004).
Consultation and Relational Empathy measure (CARE) | 4 weeks following baseline visit
  The Consultation and Relational Empathy measure (CARE) is a 10-item self-report measure of patients' experience of clinical encounters. It shows high internal reliability (Cronbach's α of 0.92) and sufficient evidence of face validity (feedback from 10 patients) and convergent validity (r = 0.85 versus Reynolds Empathy Measure (RES)) (Mercer et al., 2004).
An adaptation of the Medical Interview Satisfaction Scale (MISS-21) | 4 weeks following baseline visit
  The Medical Interview Satisfaction Scale (MISS-21) is a 21-item self-report measure of patients' satisfaction with doctor consultations, validated in British general practice populations. Internal consistency scores ranges between Cronbach's α of 0.67 and 0.92 for the four subscales. There is sufficient evidence construct validity of the MISS-21 with highly significant positive correlations (0.21-0.63) between MISS-21 scores and aspects of satisfaction with previous consultations (Meakin & Weinman, 2002). The FORECAST 2 study will make use of selected questions from MISS-21 that are relevant to the clinical encounters with therapeutic radiographers.
5 EQ-5D-3L | 6-8 weeks after treatment
  The EQ-5D-3L is a standardised instrument for use as a measure of health outcome and was developed by the EuroQol Research foundation. It consists of five questions relating to five dimensions of health; mobility, self-care, usual activities, pain and discomfort and anxiety and depression. The EQ-5D has well-established validity and reliability and has been used in many studies of patients with a variety of chronic conditions in many different countries (Schrag et al., 2000; Walters & Brazier, 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Humphris, PhD, Principal Investigator — University of St Andrews
Locations (2):
- United Kingdom (2):
  - NHS Lothian Edinburgh Cancer Centre, Edinburgh
  - University of St Andrews, St Andrews

REFERENCES:
- [Background] Crawford JR, Henry JD. The positive and negative affect schedule (PANAS): construct validity, measurement properties and normative data in a large non-clinical sample. Br J Clin Psychol. 2004 Sep;43(Pt 3):245-65. doi: 10.1348/0144665031752934. PMID 15333231
- [Background] Mercer SW, Maxwell M, Heaney D, Watt GC. The consultation and relational empathy (CARE) measure: development and preliminary validation and reliability of an empathy-based consultation process measure. Fam Pract. 2004 Dec;21(6):699-705. doi: 10.1093/fampra/cmh621. Epub 2004 Nov 4. PMID 15528286
- [Background] Meakin R, Weinman J. The 'Medical Interview Satisfaction Scale' (MISS-21) adapted for British general practice. Fam Pract. 2002 Jun;19(3):257-63. doi: 10.1093/fampra/19.3.257. PMID 11978716
- [Background] Schrag A, Selai C, Jahanshahi M, Quinn NP. The EQ-5D--a generic quality of life measure-is a useful instrument to measure quality of life in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jul;69(1):67-73. doi: 10.1136/jnnp.69.1.67. PMID 10864606
- [Background] Walters SJ, Brazier JE. Comparison of the minimally important difference for two health state utility measures: EQ-5D and SF-6D. Qual Life Res. 2005 Aug;14(6):1523-32. doi: 10.1007/s11136-004-7713-0. PMID 16110932
- [Background] Humphris GM, Watson E, Sharpe M, Ozakinci G. Unidimensional scales for fears of cancer recurrence and their psychometric properties: the FCR4 and FCR7. Health Qual Life Outcomes. 2018 Feb 9;16(1):30. doi: 10.1186/s12955-018-0850-x. PMID 29471823
- [Result] Barracliffe L, Yang Y, Cameron J, Bedi C, Humphris G. Does emotional talk vary with fears of cancer recurrence trajectory? A content analysis of interactions between women with breast cancer and their therapeutic radiographers. J Psychosom Res. 2018 Mar;106:41-48. doi: 10.1016/j.jpsychores.2018.01.004. Epub 2018 Jan 9. PMID 29455898
- [Derived] van Beusekom M, Cameron J, Bedi C, Banks E, Harris R, Humphris G. Using Co-design With Breast Cancer Patients and Radiographers to Develop "KEW" Communication Skills Training. Front Psychol. 2021 Feb 22;12:629122. doi: 10.3389/fpsyg.2021.629122. eCollection 2021. PMID 33692727
- [Derived] van Beusekom M, Cameron J, Bedi C, Banks E, Kelsey T, Humphris G. Development, acceptability and feasibility of a communication skills training package for therapeutic radiographers to reduce fear of recurrence development in breast cancer patients (FORECAST2). Pilot Feasibility Stud. 2018 Sep 18;4:148. doi: 10.1186/s40814-018-0338-9. eCollection 2018. PMID 30237899